CLINICAL TRIAL: NCT01683474
Title: Clinical Evaluation of the Safety and Performance of Percutaneous Implantation of the Venus MedTech Aortic Valve Prosthesis for Patients Who Cannot Undergo Surgical Valve Replacement
Brief Title: Safety and Performance of TAVI of Venus MedTech Aortic Valve Prosthesis
Acronym: Venus-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Venus MedTech (HangZhou) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Venus-A Study
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Calcification
Keywords: aortic valve stenosis; Calcification; TAVI; aortic valve Prosthesis
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of; Calcinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Venus A-Valve (Experimental): single arm with intervention that percutaneous implantation of the Venus MedTech Aortic Valve Prosthesis
  Interventions: Device: Venus MedTech Aortic Valve Prosthesis

INTERVENTIONS:
Device: Venus MedTech Aortic Valve Prosthesis — Percutaneous implantation of aortic valve of Venus-A
  Other Names: Venus A-Valve; Venus A-Valve System

SUMMARY:
1. objectives

   * Evaluate the performance of Venus MedTech aortic valve prosthesis intervention by femoral artery
   * Evaluate safety and clinical benefit of percutaneous implantation of the Venue MedTech aortic valve prosthesis.
   * Continuous observe 12 months of safety and efficacy.
2. Approximately 80 patients presenting with native aortic valve stenosis necessitating valve replacement which are considered unsuitable for Surgical Valve Replacement, with a high surgical risk, as attested to by both the surgeon and the cardiologist are recruited in the study.
3. Safety and performance will be evaluated at discharge and at 30 days post procedure. Valve safety, performance and placement will be followed up at 6 and 12 months post-procedure.

DETAILED DESCRIPTION:
A prospective OPC study to evaluate its performance and long-term safety and effectiveness of Venus-A aortic valve.

ELIGIBILITY:
Inclusion Criteria:

* Senile degenerative aortic valve stenosis with echocardiography derived criteria: mean gradient ≥ 40 mm Hg, or jet velocity ≥ 4.0 m/s, or an aortic valve area (AVA) of < 0.8 cm2 (or AVA index < 0.5 cm2/m2)
* Symptomatic due to aortic valve stenosis as demonstrated by NYHA Functional Class ≥ II
* The subject or the subject's legal representative was informed of the nature of the study, agreed to its provisions and provided written informed consent as approved by the Institutional Review Board of the respective clinical site.
* The subject agreed to comply follow-up evaluation
* is evaluated by at least one cardiologist and two cardiovascular surgeon, and they agreed that medical factors precluding operation suitable for surgery (the probability of death or serious, irreversible morbidity exceeded 50%)
* STS score ≥ 10%

Exclusion Criteria:

* Patient refuses aortic valve replacement surgery.
* Evidence of an acute myocardial infarction ≤ 1 month before the intended treatment [defined as: Q wave MI, or non-Q wave MI with total CK elevation of CK-MB ≥ twice normal in the presence of MB elevation and/or troponin level elevation (WHO definition)].
* Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is non-calcified.
* Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+).
* Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days （6 month if DES implant）
* Implanted any heart valve prosthesis, prosthetic valve ring, severe mitral valve ring calcification (MAC), severe（>3＋）mitral valve insufficiency, or Gorelin symptom
* Blood dyscrasia such as leukopenia (WBC < 3×109/L), acute anemia (Hgb < 90 g/L), thrombocytopenia (PLT < 50×109/L), bleeding diathesis, or history of coagulopathy.
* Untreated clinically significant coronary artery disease requiring revascularization
* Hemodynamic instability requiring inotropic therapy or mechanical hemodynamic support devices
* Need for emergency surgery for any reason
* Hypertrophic cardiomyopathy with or without obstruction (HOCM)
* Severe ventricular dysfunction with LVEF < 20%
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Active peptic ulcer or upper gastro-intestinal bleeding within the prior 3 months
* A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, Nitinol, or sensitivity to contrast media which cannot be adequately pre-medicated.
* Native aortic annulus size < 20 mm or> 29 mm as measured by echocardiogram.
* Cerebrovascular Accident (CVA) within 6 months, including TIA.
* Renal insufficiency (creatinine > 3.0 mg/dL) and/or end stage renal disease requiring chronic dialysis.
* Life expectancy < 12 months
* Significant abdominal or thoracic aorta disease, including aneurysm (defined as maximal luminal diameter 5cm or greater), marked tortuosity (hyperacute bend), aortic arch atheroma (especially if thick [> 5 mm], protruding or ulcerated), narrowing of the abdominal aorta (especially with calcification and surface irregularities), or severe "unfolding" and tortuosity of the thoracic aorta
* Iliofemoral vessel characteristics that would preclude safe placement of 16F or 18F introducer sheath such as severe obstructive calcification, severe tortuosity or vessel size diameter < 7 mm.
* Currently participating in an investigational drug or another device study.
* Active bacterial endocarditis or other active infections.
* Bulky calcified aortic valve leaflets in close proximity to coronary ostia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-02 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
All cause mortality and major stroke at 12 months post-procedure. | 12 months post-procedure

SECONDARY OUTCOMES:
Valve performance and placement at 6 and 12 months post-procedure | 6 and 12 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ruilin Gao, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fu Wai Hospital, CAMS & PUMA, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lei WH, Liao YB, Wang ZJ, Ou YW, Tsauo JY, Li YJ, Xiong TY, Zhao ZG, Wei X, Meng W, Feng Y, Chen M. Transcatheter Aortic Valve Replacement in Patients with Aortic Stenosis Having Coronary Cusp Fusion versus Mixed Cusp Fusion Nonraphe Bicuspid Aortic Valve. J Interv Cardiol. 2019 Nov 3;2019:7348964. doi: 10.1155/2019/7348964. eCollection 2019. PMID 31777470
- [Derived] Liao YB, Li YJ, Xiong TY, Ou YW, Lv WY, He JL, Li YM, Zhao ZG, Wei X, Xu YN, Feng Y, Chen M. Comparison of procedural, clinical and valve performance results of transcatheter aortic valve replacement in patients with bicuspid versus tricuspid aortic stenosis. Int J Cardiol. 2018 Mar 1;254:69-74. doi: 10.1016/j.ijcard.2017.12.013. Epub 2017 Dec 9. PMID 29246428
- [Derived] Jilaihawi H, Wu Y, Yang Y, Xu L, Chen M, Wang J, Kong X, Zhang R, Wang M, Lv B, Wang W, Xu B, Makkar RR, Sievert H, Gao R. Morphological characteristics of severe aortic stenosis in China: imaging corelab observations from the first Chinese transcatheter aortic valve trial. Catheter Cardiovasc Interv. 2015 Mar;85 Suppl 1:752-61. doi: 10.1002/ccd.25863. Epub 2015 Feb 19. PMID 25630494